CLINICAL TRIAL: NCT01190462
Title: Safety and Efficacy of the Addition of Simvastatin to Cetuximab in K-ras Mutant Advanced or Metastatic Colorectal Cancer Patients. A Single-Arm, Multicenter, Phase II Study Using a Simon Two Stage Design.
Brief Title: Cetuximab and Simvastatin in Treating Patients With Advanced or Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: DUT-LUMC-838; CDR0000683942 (Registry Identifier: PDQ (Physician Data Query)); NL-30642-058-10; EUDRACT-2009-017384-42; EU-21065
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2011-04

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Simvastatin

INTERVENTIONS:
Biological: cetuximab
Drug: simvastatin
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Simvastatin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Simvastatin may help cetuximab work better by making tumor cells more sensitive to cetuximab. Giving cetuximab together with simvastatin may kill more tumor cells.

PURPOSE: This phase II trial is studying giving cetuximab together with simvastatin in treating patients with advanced or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the percentage of patients with k-ras mutant, advanced or metastatic colorectal cancer who are free from progression and alive after 12.5 weeks following the first dose of cetuximab in combination with simvastatin.

Secondary

* To determine the correlation between overall response rate, progression-free survival, overall survival, and safety with skin toxicity and efficacy.
* To determine the predictive value of PTEN, PIK3CA, b-raf, and ERK and MEK status. (exploratory)
* To determine the predictive value of SNPs, proteomics, and circulating DNA. (exploratory)
* To evaluate cholesterol, proteomics, and circulating DNA as biomarkers in this setting. (exploratory)

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV weekly and oral simvastatin once daily on days 1-7. Courses repeat every 7 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected for laboratory studies at baseline, during study, and after completion of study.

After completion of study therapy, patients are followed up for 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of advanced or metastatic colorectal cancer
* Progressive disease in the past 3 months
* Failed prior oxaliplatin-, fluorouracil (5-FU)-, and irinotecan-containing regimens AND have the presence of a k-ras mutation within codon 12, 13, or 61

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Adequate organ function
* No history of toxicity during statin use
* No other malignancy within the past 5 years
* No history of severe pulmonary disease
* No clinically relevant coronary artery disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior epidermal growth factor receptor (EGFR)-targeting agents
* No concurrent verapamil or amiodarone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients free from progression and alive after 12.5 weeks following the first dose of treatment

SECONDARY OUTCOMES:
Correlation between overall response rate, progression-free survival, overall survival, and safety with skin toxicity and efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gelderblom, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Amphia Ziekenhuis - locatie Langendijk, Breda
  - Leiden University Medical Center, Leiden